CLINICAL TRIAL: NCT02859987
Title: Randomized Controlled Trial of Ultrasound-guided Versus Landmark Technique for Peripherally Inserted Central Catheter (PICC) Placement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Equipo de Terapia Intravenosa (Other)
Collaborators: Hospital San Carlos, Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ETI-HCSC-01
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: PICC Placement
Keywords: US; Nursing Services
MeSH Terms: interventions — Ultrasonography

ARMS (2):
- Landmark Technique (Active Comparator): Blinded method for catheter placement
  Interventions: Procedure: PICC Placement by Landmark Technique
- Ultrasound-guided Technique (Experimental): Use sonography for catheter placement
  Interventions: Procedure: PICC Placement by Ultrasound-guided Technique; Device: Ultrasound Scan

INTERVENTIONS:
Procedure: PICC Placement by Landmark Technique — Comparison of two different techniques for PICC Placement (Landmark versus Ultrasound-guided)
  Arms: Landmark Technique
Procedure: PICC Placement by Ultrasound-guided Technique — Comparison of two different techniques for PICC Placement (Landmark versus Ultrasound-guided)
  Arms: Ultrasound-guided Technique
Device: Ultrasound Scan — Initially the nurses use ultrasound for explore venous anatomy and then they use real-time ultrasound imaging during needle placement
  Arms: Ultrasound-guided Technique

SUMMARY:
Peripherally Inserted Central Catheter (PICC) are intravascular devices used on patients undergoing IV therapy. Insertion of these catheters can be achieved either by using the anatomical landmarks for the veins or using ultrasound guidance. The guidelines recommend the use of ultrasound guidance for central venous access catheterization to facilitate central venous cannulation (CVC) and to reduce the risk of complications, but the scientific evidence is limited and heterogeneous.

This is a prospective randomized clinical trial in adults patients requiring peripherally inserted central catheter (PICC) placement for intravenous therapy.

The principal aim of this randomized clinical trial is to evaluate the effectiveness of ultrasound-guidance technique for successfully peripherally central venous catheterisation in the first attempt versus landmark method, in the context of PICC cannulation.

Patients are randomized (1:1) in two groups: Control arm (landmark technique) versus Experimental group (ultrasound guidance technique). In order to avoid expected biases the investigators stratified the cases by difficulty for venous cannulation. Crossover was allowed if catheterisation could not be reached after two unsuccessful venipunctures, to prevent suffering of the patients and troubles in its care.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Patients with indication of PICC insertion for long-term intravenous therapy

Exclusion Criteria:

* Peripheral vascular disease
* Injecting drug users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evidence of catheter inserted at first attempt, correctly located (after chest X-ray performed) and proper working, confirmed by the nurse | Within the first 6 hours after placement
  The principal aim is to evaluate the effectiveness of ultrasound-guidance technique for successfully peripherally central venous catheterisation in the first attempt versus landmark method, in the context of PICC cannulation

CONTACTS AND LOCATIONS:
Overall Officials: Maria Montealegre, RN, IV Nurse, Study Director — Hospital Universitario Clinico San Carlos